CLINICAL TRIAL: NCT06879093
Title: Adaptation Plan for Culturally Competent Care (PAACI) in the Acute Psychiatric Unit.
Acronym: PAACI
Status: Active, not recruiting | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Amira Trabsa, Psychiatrist and coordinator of the psychiatric acute unit., Hospital del Mar
Other Study IDs: 2021/10025
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Mental Disorders; Cultural Competency; Psychiatric Hospitalization
Keywords: Cultural Competence; Mental Health Equity; Psychiatric Care; Immigrant Health; Acute Psychiatric Unit; Cross-Cultural Psychiatry; Health Disparities
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Immigrant patients in acute psychiatric unit: This cohort includes immigrant patients admitted to the Acute Psychiatric Unit at Parc de Salut Mar. The study will analyze key clinical indicators before and after the implementation of the Adaptation plan for culturally competent care (PAACI) to assess its impact on patient outcomes.

SUMMARY:
This observational study aims to design, implement, and evaluate the Adaptation Plan for Culturally Competent Care (PAACI) in the Acute Psychiatric Unit of Parc de Salut Mar, Barcelona. The study focuses on improving healthcare quality for immigrant patients by reducing cultural and linguistic barriers in psychiatric care.

The PAACI program includes educational materials in multiple languages, enhanced collaboration with social services, training for healthcare professionals in cultural competence, and the use of interpretation devices. Key outcomes include reducing mechanical restraints, improving patient adherence to treatment, decreasing hospital readmissions, and increasing outpatient care engagement.

The study will analyze data from immigrant patients admitted to the Acute Psychiatric Unit one year before and after the implementation of PAACI, using various clinical and patient satisfaction indicators. This initiative aims to promote equal and equitable healthcare for diverse populations, potentially serving as a model for other mental health units.

DETAILED DESCRIPTION:
This study evaluates the implementation of the Adaptation Plan for Culturally Competent Care (PAACI) in an Acute Psychiatric Unit. The project aims to improve psychiatric care for immigrant patients by addressing cultural and linguistic barriers.

The study follows an observational design, comparing key clinical outcomes before and after the PAACI implementation. It includes measures such as staff training in cultural competence, improved coordination with social and healthcare services, and the introduction of multilingual patient education materials.

The primary focus is on enhancing healthcare equity, reducing the use of mechanical restraints, improving patient adherence to outpatient care, and decreasing hospital readmissions. Findings from this study may inform future adaptations of culturally competent care models in psychiatric settings.

ELIGIBILITY:
Inclusion Criteria:

* immigrant patients admitted to the acute psychiatric unit
* age 18 or older
* hospitalization during the study period (12 months post-paaci implementation)

Exclusion Criteria:

* patients with severe cognitive impairment preventing informed consent
* individuals with acute medical conditions requiring transfer to another service
* refusal to participate or withdraw consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: this study focuses on immigrant patients admitted to the acute psychiatric unit at hospital del mar. participants will be individuals aged 18 or older who experience acute mental health crises requiring hospitalization. the study will analyze clinical outcomes before and after the implementation of the paaci program, which aims to improve culturally competent psychiatric care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
reduction in mechanical restraints | 12 months after paaci implementation
  this measure evaluates the impact of the paaci program on the total number of mechanical restraints used in immigrant patients admitted to the acute psychiatric unit. data will be compared before and after program implementation.

SECONDARY OUTCOMES:
Hospital Readmission Rate Among Immigrant Patients | 12 months after paaci implementation
  Comparison of the number of readmissions within 30 days post-discharge among immigrant patients before and after PAACI implementation.
Length of Hospital Stay for Immigrant Patients | 12 months after PAACI implementation
  Evaluation of the average length of hospitalization for immigrant patients before and after PAACI implementation.
Patient adherence to outpatient mental health services | 12 months after PAACI implementation
  Assessment of the percentage of discharged immigrant patients who attend their first outpatient follow-up appointment after hospitalization.
patient and staff satisfaction levels | 12 months after paaci implementation
  comparison of patient and staff satisfaction levels with psychiatric care before and after paaci implementation, using validated survey tools.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar-Centro Forum, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to confidentiality considerations and ethical regulations. The study focuses on evaluating a healthcare intervention rather than collecting individualized clinical data for external research purposes. all collected data will be analyzed in aggregate form to ensure participant privacy and compliance with data protection laws.

REFERENCES:
- [Background] Elwell-Sutton TM, Jiang CQ, Zhang WS, Cheng KK, Lam TH, Leung GM, Schooling CM. Inequality and inequity in access to health care and treatment for chronic conditions in China: the Guangzhou Biobank Cohort Study. Health Policy Plan. 2013 Aug;28(5):467-79. doi: 10.1093/heapol/czs077. Epub 2012 Sep 16. PMID 22987824
- [Background] Pereira ME, Alvaro Estramiana JL, Schweiger Gallo I. Essentialism and the expression of social stereotypes: a comparative study of Spain, Brasil and England. Span J Psychol. 2010 Nov;13(2):808-17. doi: 10.1017/s1138741600002468. PMID 20977029
- [Background] Dein S. ABC of mental health. Mental health in a multiethnic society. BMJ. 1997 Aug 23;315(7106):473-6. doi: 10.1136/bmj.315.7106.473. No abstract available. PMID 9284670
- [Background] Bhui K, Warfa N, Edonya P, McKenzie K, Bhugra D. Cultural competence in mental health care: a review of model evaluations. BMC Health Serv Res. 2007 Jan 31;7:15. doi: 10.1186/1472-6963-7-15. PMID 17266765
- [Background] Betancourt TS, Newnham EA, Birman D, Lee R, Ellis BH, Layne CM. Comparing Trauma Exposure, Mental Health Needs, and Service Utilization Across Clinical Samples of Refugee, Immigrant, and U.S.-Origin Children. J Trauma Stress. 2017 Jun;30(3):209-218. doi: 10.1002/jts.22186. Epub 2017 Jun 6. PMID 28585740